CLINICAL TRIAL: NCT01137474
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Dapagliflozin in Subjects With Type 2 Diabetes With Inadequately Controlled Hypertension on an Angiotensin-Converting Enzyme Inhibitor (ACEI) or Angiotensin Receptor Blocker (ARB)
Brief Title: A Study of BMS-512148 (Dapagliflozin) in Patients With Type 2 Diabetes and Inadequately Controlled Hypertension on an Angiotensin-Converting Enzyme Inhibitor or Angiotensin Receptor Blocker
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB102-073 ST; 2010-019797-32 (EudraCT Number)
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases; Angiotensin Receptor Antagonists; Angiotensin-Converting Enzyme Inhibitors; Hypoglycemic Agents; Pharmacologic Actions; Physiological Effects of Drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dapagliflozin, 10 mg (Experimental): Oral tablets administered as 10 mg once daily for up to 12 weeks
  Interventions: Drug: Dapagliflozin
- Placebo-matching dapagliflozin (Placebo Comparator): Oral tablets administered once daily in the morning
  Interventions: Drug: Placebo-matching dapagliflozin
- Dapagliflozin, 2. 5 mg (Experimental): Oral tablets administered as 2.5 mg once daily for up to 12 weeks (Arm discontinued as of Protocol Amendment 8)
  Interventions: Drug: Dapagliflozin
- Dapagliflozin, 5 mg (Experimental): Oral tablets administered as 5 mg once daily for up to 12 weeks (Arm discontinued as of Protocol Amendment 8)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Oral tablets administered as 2.5, 5, or 10 mg, once daily for up to 12 weeks
  Other Names: BMS-512148
  Arms: Dapagliflozin, 10 mg; Dapagliflozin, 2. 5 mg; Dapagliflozin, 5 mg
Drug: Placebo-matching dapagliflozin — Oral tablets administered as 0 mg once daily for up to 12 weeks
  Arms: Placebo-matching dapagliflozin

SUMMARY:
The purpose of this study is to learn whether dapagliflozin, after 12 weeks, can improve (decrease) blood pressure in patients with type 2 diabetes with uncontrolled hypertension who are on an angiotensin-converting enzyme inhibitor or an angiotensin receptor blocker. The safety of this treatment will also be studied.

ELIGIBILITY:
Key inclusion criteria

* Participants willing and able to give signed and written informed consent
* Males and females, aged 18 to 89 years, who have type 2 diabetes with inadequate glycemic control (hemoglobin A1c between 7% and 10.5%) and uncontrolled hypertension (seated systolic blood pressure of 140 to 165 mm Hg and seated diastolic blood pressure 85 to 105 mm Hg)
* Mean 24-hour BP>=130/80 mmHg determined by ABPM
* Stable dose of oral antidiabetic agent (OAD) for at least 6 weeks (12 weeks for thiazolidinedione) or a stable daily dose of insulin as monotherapy or in combination with another OAD, for 8 weeks, and a stable dose of an angiotensin-converting enzyme inhibitor or angiotensin-receptor blocker for at least 4 weeks
* C-peptide level ≥0.8 ng/mL
* Body mass index ≤ 45.0 kg/m^2

Key exclusion criteria

* Aspartate aminotransferase or alanine aminotransferase level >3*upper limit of normal (ULN)
* Serum total bilirubin level >1.5*ULN
* Serum creatinine ≥2.0 mg/dL unless subject was on metformin, where exclusionary limits were serum creatinine ≥1.50 mg/dL for men and ≥1.40 mg/dL for women
* Estimated creatinine clearance of <60 mL/min
* Hemoglobin ≤10.0 g/dL for men and ≤9.0 g/dL for women
* Creatine kinase >3*ULN
* Positive for hepatitis B surface antigen
* Positive for antihepatitis C virus antibody
* Abnormal free T4 value
* History of diabetes insipidus
* Symptoms of poorly controlled diabetes that would preclude participation in this trial, including but not limited to, marked polyuria and polydipsia with greater than 10% weight loss during the 3 months prior to enrollment.
* History of diabetic ketoacidosis or hyperosmolar nonketotic coma
* History of malignant and accelerated hypertension
* Known or suspected secondary hypertension
* Any of the following within 6 months of enrollment visit:

  * Myocardial infarction
  * Cardiac surgery or revascularization (coronary artery bypass surgery /percutaneous transluminal coronary angioplasty)
  * Unstable angina
  * Unstable congestive heart disease or New York Heart Association Class III or IV
  * Transient ischemic attack or significant cerebrovascular disease
  * Unstable or previously undiagnosed arrhythmia

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2996 (Actual)
Dates: Start 2010-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (292):
- United States (164):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Horizon Research Group, Inc., Mobile, Alabama
  - Iicr, Inc. (International Institute Of Clinical Research), Ozark, Alabama
  - Hope Research Institute, Phoenix, Arizona
  - 43rd Medical Associates, Phoenix, Arizona
  - Central Phoenix Medical Clinic, Llc, Tempe, Arizona
  - Clinical Research Advantage/Desert Clinical Research, Tempe, Arizona
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Aureus Research, Inc., Little Rock, Arkansas
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Orange County Research Institute, Anaheim, California
  - Cmp Research, Anaheim, California
  - Med Center, Carmichael, California
  - Catalina Research Institute, Llc, Chino, California
  - Southland Clinical Research Center, Inc., Fountain Valley, California
  - Marin Endocrine Care & Research, Inc., Greenbrae, California
  - Del Rosario Medical Clinic, Inc., Huntington Park, California
  - Time Clinical Research Inc., Huntington Park, California
  - Marina Raikhel, M.D., F.A.A.F.P, Lomita, California
  - Clinica Medica San Miguel, Los Angeles, California
  - American Institute Of Research, Los Angeles, California
  - Randall G. Shue, D.O., Los Angeles, California
  - National Research Inst, Los Angeles, California
  - Quest Diagnostics West Hills, Los Angeles, California
  - Diabetes Medical Center Of California, Northridge, California
  - Valley Clinical Trials, Northridge, California
  - Lucita M. Cruz,Md.,Inc., Norwalk, California
  - Sds Clinical Trials, Orange, California
  - Integrated Research Group, Inc., Riverside, California
  - Quality Control Research, Inc, Sacramento, California
  - Crest Clinical Trials, Inc., Santa Ana, California
  - Orrin M. Troum, Md And Medical Associates, Santa Monica, California
  - Orange County Research Center, Tustin, California
  - University Clinical Investigators, Inc., Tustin, California
  - Infosphere Clinical Research, Inc., West Hills, California
  - Aurora Family Medicine, P.C., Aurora, Colorado
  - Horizons Clinical Research Center, Llc, Denver, Colorado
  - Chase Medical Research, Llc, Waterbury, Connecticut
  - Zasa Clinical Research, Boynton Beach, Florida
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Meridien Research, Brooksville, Florida
  - Family Care Associates Of Nw Fl, Chipley, Florida
  - Innovative Research Of West Florida, Inc, Clearwater, Florida
  - Clinical Research Of South Florida, Coral Gables, Florida
  - Avail Clinical Research, Llc, DeLand, Florida
  - In Vivo Clinical Research, Doral, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - The Community Research Of South Florida, Hialeah, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Flcri Global Research, Llc, Miami, Florida
  - International Research Associates, Llc, Miami, Florida
  - Clinical Research Of Miami, Inc., Miami, Florida
  - Apf Research, Llc, Miami, Florida
  - Community Research Foundation, Inc., Miami, Florida
  - Medical Research Marseilles, Miami, Florida
  - Baptist Diabetes Associates, Pa, Miami, Florida
  - Newphase Clinical Trials, Inc., Miami Beach, Florida
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Compass Research, Llc, Orlando, Florida
  - Florida Institute For Clinical Research, Llc, Orlando, Florida
  - South Miami Clinical Research, Llc, South Miami, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Perimeter Institute For Clinical Research, Atlanta, Georgia
  - Bainbridge Medical Associates, Bainbridge, Georgia
  - River Birch Research Alliance, Llc, Blue Ridge, Georgia
  - In-Quest Medical Research, Llc, Duluth, Georgia
  - Middle Georgia Clinical Research Center, Llc, Perry, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - James R. Herron, Md, Ltd, Chicago, Illinois
  - So. Illinois Clin Res Ctr @ Div Of Kevin L Pritchett Md, Pc, O'Fallon, Illinois
  - Springfield Diabetes And Endocrine Center, Springfield, Illinois
  - American Health Network Of Indiana Llc, Avon, Indiana
  - Investigators Research Group, Llc, Brownsburg, Indiana
  - American Health Network Of In Llc, Franklin, Indiana
  - Laporte County Institute For Clinical Research, Inc., Michigan City, Indiana
  - American Health Network Of In Llc, Muncie, Indiana
  - Medical Development Centers, Llc, Baton Rouge, Louisiana
  - Crescent City Clinical Research Center, Metairie, Louisiana
  - Acadia Clinical Research, Llc, Bangor, Maine
  - Alternative Primary Care, Silver Spring, Maryland
  - Neurocare, Inc., Brookline, Massachusetts
  - Genesis Clinical Research, Llc, Fall River, Massachusetts
  - Hci-Metromedic Walk-In Medical Office, New Bedford, Massachusetts
  - Atlantic Clinical Trials, Llc, Watertown, Massachusetts
  - Providence Park Clinical Research, Novi, Michigan
  - The Center For Clinical Trials, Biloxi, Mississippi
  - Phillips Medical Services, Pllc, Jackson, Mississippi
  - Jackson Clinic, Rolling Fork, Mississippi
  - Jefferson City Medical Group, Jefferson City, Missouri
  - St. Louis Center For Clinical Research, St Louis, Missouri
  - Kcumb Dybedal Clinical Research Center, Kansas City, Montana
  - Clin Research Advantage, Inc. James Meli, Do Family Pracice, Henderson, Nevada
  - Office Of Ted Thorp, Md, Las Vegas, Nevada
  - Independent Clinical Researchers@ Wolfson Medical Center, Las Vegas, Nevada
  - Clinical Research Advantage, Inc., Las Vegas, Nevada
  - Palm Medical Research Center, Las Vegas, Nevada
  - Joslin Diabetes Center Affiliate Of Snhmc, Nashua, New Hampshire
  - Central Jersey Medical Research Center, Elizabeth, New Jersey
  - Premier Research, Trenton, New Jersey
  - Medex Healthcare Research, Inc., New York, New York
  - Digiovanna Institute For Medical Education & Research, North Massapequa, New York
  - Southgate Medical Group, West Seneca, New York
  - Barat Research Group, Inc., Charlotte, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Pmg Research Of Wilmington Llc, Wilmington, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Community Health Care, Inc., Canal Fulton, Ohio
  - Community Research, Cincinnati, Ohio
  - Cleveland Sleep Research Center, Middleburg Heights, Ohio
  - Clinical Research Source, Inc, Perrysburg, Ohio
  - Integris Family Care Central, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Integris Family Care Yukon, Yukon, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Fanno Creek Clinic, Portland, Oregon
  - Southeastern Pa Medical Institute, Broomall, Pennsylvania
  - Abington Memorial Hos/Feasterville Family Health Care Center, Feasterville-Trevose, Pennsylvania
  - The Clinical Trial Center, Llc, Jenkintown, Pennsylvania
  - Arcuri Clinical Research Llc, Philadelphia, Pennsylvania
  - Philadelphia Health Associates - Adult Medicine, Philadelphia, Pennsylvania
  - Banksville Medical Pc, Pittsburgh, Pennsylvania
  - Research Across America, Reading, Pennsylvania
  - Pish Medical Associates, Uniontown, Pennsylvania
  - Greater Providence Clinical Research, Llc, Warwick, Rhode Island
  - Southeastern Research Associates, Inc., Anderson, South Carolina
  - Southeastern Research Associates, Inc., Greenville, South Carolina
  - Hillcrest Clinical Reseach, Llc, Simpsonville, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Chattanooga Research & Medicine, Pllc, Chattanooga, Tennessee
  - Complete Family Care Of Knoxville, Pllc, Knoxville, Tennessee
  - Premier Internal Medicine, Memphis, Tennessee
  - Arlington Family Research Center, Inc., Arlington, Texas
  - Krk Medical Research, Dallas, Texas
  - Research Institute Of Dallas, Dallas, Texas
  - Internal Medicine Clinical Research, Dallas, Texas
  - Renaissance Clinical Research And Hypertension Pllc, Dallas, Texas
  - Sergio F. Rovner, M.D., El Paso, Texas
  - Mercury Clinical Research, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Excel Clinical Research, Llc, Houston, Texas
  - Lone Star Clinical Research, Houston, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - North Hills Medical Research, Inc., North Richland Hills, Texas
  - Med-Olam Clinical Research, Pasadena, Texas
  - Lisa E. Medwedeff, Md, Pa, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Abbott Clinical Research Group, Inc., San Antonio, Texas
  - Covenant Clinical Research, Pa, San Antonio, Texas
  - Breco Research, Ltd, Sugarland, Texas
  - Pioneer Research Solutions, Inc., Sugarland, Texas
  - Exodus Healthcare Network, Magna, Utah
  - Wasatch Endocrinology And Diabetes Specialists, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Millennium Clinical Trials Llc, Arlington, Virginia
  - Burke Internal Medicine And Research, Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Hampton Roads Center For Clinical Research, Inc., Suffolk, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Sound Medical Research, Port Orchard, Washington
- Canada (6):
  - Local Institution, Kelowona, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Brampton, Ontario
  - Local Institution, Granby, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Colombia (6):
  - Local Institution, Medellín, Antioquia
  - Local Institution, Bogota, Cundinamarca
  - Local Institution, Armenia, Quindío Department
  - Local Institution, Cali, Valle del Cauca Department
  - Local Institution, Barranquilla
  - Local Institution, Bogotá
- Czechia (6):
  - Local Institution, Beroun
  - Local Institution, Cheb
  - Local Institution, Havířov
  - Local Institution, Liberec
  - Local Institution, Ostrava
  - Local Institution, Prague
- Denmark (3):
  - Local Institution, Copenhagen
  - Local Institution, Frederiksberg
  - Local Institution, Slagelse
- Finland (2):
  - Local Institution, Kokkola
  - Local Institution, Oulu
- Germany (15):
  - Local Institution, Aschaffenburg, Bavaria
  - Local Institution, Vellmar, Hesse
  - Local Institution, Duisburg, North Rhine-Westphalia
  - Local Institution, Bad Kreuznach
  - Local Institution, Berlin
  - Local Institution, Karlsruhe
  - Local Institution, Köthen
  - Local Institution, Kronshagen
  - Local Institution, Langenfeld
  - Local Institution, Lüneburg
  - Local Institution, Magdeburg
  - Local Institution, Mainz
  - Local Institution, Mannheim
  - Local Institution, Pirna
  - Local Institution, Saarbrücken
- Hungary (11):
  - Local Institution, Gyöngyös, Heves County
  - Local Institution, Eger
  - Local Institution, Hatvan
  - Local Institution, Miskolc
  - Local Institution, Nagykanizsa
  - Local Institution, Nyíregyháza
  - Local Institution, Sátoraljaújhely
  - Local Institution, Sopron
  - Local Institution, Szeged
  - Local Institution, Szekszárd
  - Local Institution, Szentes
- India (15):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Vijayawada, Andhra Pradesh
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Belagavi, Karnatka
  - Local Institution, Indore, Madhya Pradesh
  - Local Institution, Nagpur, Maharashtra
  - Local Institution, New Delhi, National Capital Territory of Delhi
  - Local Institution, Delhi, New Delhi
  - Local Institution, Jaipur, Rajasthan
  - Local Institution, Coimbatore, Tamil Nadu
  - Local Institution, Madurai, Tamil Nadu
  - Local Institution, Bangalore
  - Local Institution, Hyderabad
  - Local Institution, Manipal
  - Local Institution, Nagpur
- Mexico (15):
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Torreón, Coahuila
  - Local Institution, Durango, Durango
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Del. Benito Juarez, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Tlalpan, Mexico City
  - Local Institution, Cuautla, Morelos
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Puebla City, Puebla
  - Local Institution, Querétaro City, Querétaro
  - Local Institution, Culiacán, Sinaloa
  - Local Institution, Veracruz, Veracruz
  - Local Institution, Mérida, Yucatán
  - Local Institution, Guadalajara
- Peru (7):
  - Local Institution, Arequipa, Arequipa
  - Local Institution, Cusco, Departamento de Cusco
  - Local Institution, Ica, Ica
  - Local Institution, Chiclayo, Lambayeque
  - Local Institution, Lima, Lima Province
  - Local Institution, Lince, Lima region
  - Local Institution, Piura, Piura
- Poland (17):
  - Local Institution, Bialystok
  - Local Institution, Bydgoszcz
  - Local Institution, Chrzanów
  - Local Institution, Gdansk
  - Local Institution, Gdynia
  - Local Institution, Golub-Dobrzyń
  - Local Institution, Kamieniec Ząbkowicki
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Ostróda
  - Local Institution, Poznan
  - Local Institution, Szczecin
  - Local Institution, Warsaw
  - Local Institution, Wroc#Aw
  - Local Institution, WrocB Aw
  - Local Institution, Zamość
- Puerto Rico (3):
  - Local Institution, Cidra
  - Local Institution, Ponce
  - Local Institution, San Juan
- Romania (9):
  - Local Institution, Oradea, Bihor County
  - Local Institution, Oradea, Jud. Bihor
  - Local Institution, Timișoara, Jud. Timis
  - Local Institution, Târgu Mureş, Mureș County
  - Local Institution, Ploieşti, Prahova
  - Local Institution, Satu Mare, Satu Mare County
  - Local Institution, Sibiu, Sibiu County
  - Local Institution, Timișoara, Timiș County
  - Local Institution, Bucharest
- Russia (9):
  - Local Institution, Dzerzhinskiy
  - Local Institution, Krasnoyarsk
  - Local Institution, Moscow
  - Local Institution, Novosibirsk
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Smolensk
  - Local Institution, Yaroslavl
  - Local Institution, Yaroslav
- Spain (4):
  - Local Institution, Santiago de Compostela, A Coruna
  - Local Institution, Barcelona
  - Local Institution, La Roca del Vallès
  - Local Institution, Peralada

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- See also: Redacted_Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3669&filename=MB102073_CSP_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was originally designed with 2 additional double-blind treatment arms, dapagliflozin 2.5 and
  5 mg, but randomization of new patients into these arms stopped with implementation of Protocol Amendment 8
  on 1-11-11. Patients randomized to dapagliflozin 2.5 or 5 mg remained on their blinded medication until study completion.
Pre-assignment Details: Of 2996 participants enrolled, 944 were randomized and received double-blind treatment.
Groups:
- Placebo: Participants with type 2 diabetes and inadequate glycemic and hypertension control while taking an oral antidiabetic drug (OAD) with or without insulin and an angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB), received dapagliflozin-matching placebo daily with a morning meal.
- Dapagliflozin, 2.5 mg (Randomized Before Protocol Amendment 8): Participants with type 2 diabetes and inadequate glycemic and hypertension control while taking an OAD with or without insulin and an ACE inhibitor or ARB, received dapagliflozin, 2.5 mg, daily with a morning meal.
- Dapagliflozin, 5 mg (Randomized Before Protocol Amendment 8): Participants with type 2 diabetes and inadequate glycemic and hypertension control while taking an OAD with or without insulin and an ACE inhibitor or ARB, received dapagliflozin, 5 mg, daily with a morning meal.
- Dapagliflozin 10 mg: Participants with type 2 diabetes and inadequate glycemic and hypertension control while taking an OAD with or without insulin and an ACE inhibitor or ARB, received dapagliflozin, 10 mg, daily with a morning meal.
Period: Overall Study
Arm/Group | Placebo | Dapagliflozin, 2.5 mg (Randomized Before Protocol Amendment 8) | Dapagliflozin, 5 mg (Randomized Before Protocol Amendment 8) | Dapagliflozin 10 mg
Started | 311 | 166 | 165 | 302
Received Treatment | 311 | 166 | 165 | 302
Completed | 287 | 154 | 158 | 281
Not Completed | 24 | 12 | 7 | 21
Not completed — Adverse Event | 3 | 5 | 1 | 3
Not completed — Withdrawal by Subject | 7 | 2 | 6 | 9
Not completed — No longer met study criteria | 6 | 1 | 0 | 5
Not completed — Lost to Follow-up | 5 | 1 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2
Not completed — Other | 3 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Administrative reason by sponsor | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received a least 1 dose of double-blind study medication
Groups:
- Dapagliflozin, 2.5 mg (Randomized Before Protocol Amendment 8): Participants with type 2 diabetes and inadequate glycemic control while taking an OAD with or without insulin and an ACE inhibitor or ARB, received dapagliflozin, 2.5 mg, daily with a morning meal.
- Dapagliflozin, 5 mg (Randomized Before Protocol Amendment 8): Participants with type 2 diabetes and inadequate glycemic control while taking an OAD with or without insulin and an ACE inhibitor or ARB, received dapagliflozin, 5 mg, daily with a morning meal.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin, 2.5 mg (Randomized Before Protocol Amendment 8) | Dapagliflozin, 5 mg (Randomized Before Protocol Amendment 8) | Dapagliflozin 10 mg | Total
Number analyzed (Participants) | 311 | 166 | 165 | 302 | 944
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 259 | 141 | 142 | 260 | 802
  65 years and older to younger than 75 years | 46 | 25 | 21 | 42 | 134
  75 years and older | 6 | 0 | 2 | 0 | 8
Gender [Count of Participants; unit: Participants]
  Female | 140 | 76 | 76 | 123 | 415
  Male | 171 | 90 | 89 | 179 | 529
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 241 | 105 | 108 | 239 | 693
  Black or African American | 14 | 11 | 8 | 12 | 45
  Asian | 54 | 49 | 49 | 49 | 201
  Other | 2 | 1 | 0 | 2 | 5
Body Mass Index [Number; unit: Participants]
  Less than 25 kg/m^2 | 28 | 20 | 18 | 34 | 100
  25 kg/m^2 to 30 kg/m^2 | 131 | 67 | 63 | 95 | 356
  30 kg/m^2 and greater | 152 | 79 | 84 | 173 | 488

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Seated Systolic Blood Pressure (BP) at Week 12
Description: Seated BP was to be measured at every visit. Data after rescue medication was excluded. The patient first rested for at least 10 minutes in the seated position. Seated blood BP was determined from the mean of 3 replicated measurements obtained at least 1 minute apart. However, if the 3 consecutive seated BP readings were not within 8 mm Hg of each other, an additional 2 BP readings were to be obtained (total=5) and incorporated into the calculated mean for systolic BP and diastolic BP. For the initial BP recording, BP was measured in both arms. If the BP was higher in 1 arm, that arm was used for BP measurement. If there was no difference in BP measurements between arms, the dominant arm was used for all future BP measurements. All randomized participants who received at least 1 dose of study drug and who had nonmissing baseline and at least 1 postbaseline value during the double-blind treatment period were used for analysis. SD=standard deviation.
Time Frame: From Baseline to Week 12
Population: This study originally had 2 additional arms-dapagliflozin 2.5 and 5 mg-but randomization to these arms stopped when Protocol Amendment 8 (1-11-11) was implemented. Because endpoints focused only on 10-mg and placebo data, only patients in these arms who received study drug and who had nonmissing baseline and Week 12 values were included.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 280 | 279
mm Hg | -10.40 (0.8822) | -7.34 (0.8812)
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Change from baseline to week 12 calculated using a longitudinal repeated measures analysis using direct likelihood with fixed categorical effects of treatment, week, treatment-by-week interaction, and randomization strata and continuous fixed covariates of baseline value and baseline value by week interaction. Data after rescue were not included in the analysis. With 253 patients per group, there is >80% power to detect a difference of 3.5 mm Hg at alpha=0.05, assuming a common SD of 14 mm Hg; Test type: Superiority or Other; p = 0.0010, Longitudinal repeated measures analysis — Endpoint tested following a sequential testing procedure at two-sided alpha=0.05 to control the family-wise Type I error rate related to primary and secondary efficacy endpoints. Test performed since previous tests were significant; Only Week 12 data are presented; data from all weeks in double-blind period were included in the longitudinal repeated measures model; Mean Difference (Final Values) = -3.05, 95% CI 2-sided [-4.87 to -1.24], Standard Error of Mean 0.9251

2. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin (HbA1c) at Week 12
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. All randomized participants who received at least 1 dose of study drug and who had nonmissing baseline and at least 1 postbaseline value during the double-blind treatment period were used for analysis. SD=standard deviation.
Time Frame: From Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Dapagliflozin 10 mg
Number analyzed (Participants) | 279 | 278
Percent | -0.10 (0.0631) | -0.56 (0.0633)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Change from baseline to week 12 was calculated using a longitudinal repeated measures analysis using direct likelihood with fixed categorical effects of treatment, week, treatment-by-week interaction, and randomization strata and continuous fixed covariates of baseline value and baseline value by week interaction. With 253 subjects per group, there is >98% power to detect a difference of 0.4% at a=0.05, assuming a common SD of 1.1%; Test type: Superiority or Other; p < 0.0001, Longitudinal repeated measures analysis — [p-value comment as in outcome 1, analysis 1]; Only Week 12 data are presented; data from all weeks in the double-blind treatment period were included in the longitudinal repeated measures model; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.59 to -0.33], Standard Error of Mean 0.0673

3. Secondary Outcome: Adjusted Mean Change From Baseline in 24-Hour Ambulatory Systolic Blood Pressure at Week 12 (Last Observation Carried Forward)
Description: Ambulatory blood pressure monitoring was performed twice during the study, at baseline and at the end of study, for a duration of 24-hrs each time. If the patient met the criteria for rescue due to hypertension, a second monitoring was performed prior to the first dose of rescue medication. Initiation of the 24-hr ambulatory blood pressure monitoring began between 6 and 11 am to ensure trough blood pressure measurements were obtained. Patients were instructed to withhold all medication on the morning of the study visit and to bring their medications to the visit with them.
Time Frame: From Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Dapagliflozin 10 mg
Number analyzed (Participants) | 263 | 267
mm Hg | -6.73 (1.2427) | -9.62 (1.2277)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Change from baseline to week 12 LOCF was calculated using an ANCOVA model with treatment group as an effect and baseline value and randomization strata as covariate. Data after rescue are excluded from blood pressure analyses; Test type: Superiority or Other; p = 0.0043, ANCOVA — Endpoint tested following a sequential testing procedure at 2-sided alpha=0.05 to control the family-wise Type I error rate related to primary and secondary efficacy endpoints. Test performed since previous tests were significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.89, 95% CI 2-sided [-4.88 to -0.91], Standard Error of Mean 1.0091

4. Secondary Outcome: Adjusted Mean Change From Baseline in Seated Diastolic Blood Pressure at Week 12
Description: All randomized participants who received at least 1 dose of study drug and who had nonmissing baseline and at least 1 postbaseline value during the double-blind treatment period were used for analysis.
Time Frame: From Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Dapagliflozin 10 mg
Number analyzed (Participants) | 279 | 280
mm Hg | -4.79 (0.5418) | -5.79 (0.5425)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Change from baseline to week 12 was calculated using a longitudinal repeated measures analysis using direct likelihood with fixed categorical effects of treatment, week, treatment-by-week interaction, and randomization strata and continuous fixed covariates of baseline value and baseline value by week interaction. Data after rescue were not included in the analysis; Test type: Superiority or Other; p = 0.0843, Longitudinal repeated measures analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-2.15 to 0.14], Standard Error of Mean 0.5811

5. Secondary Outcome: Adjusted Mean Change in 24-Hour Ambulatory Diastolic Blood Pressure at Week 12 (Last Observation Carried Forward [LOCF])
Description: Ambulatory blood pressure monitoring was performed twice during the study, at baseline and at the end of study, for a duration of 24 hours each time. If the patient met the criteria for rescue due to hypertension, a second monitoring was performed prior to the first dose of rescue medication. Initiation of the 24-hour ambulatory blood pressure monitoring began between 6 and 11 am to ensure trough blood pressure measurements were obtained. Patients were instructed to withhold all medication on the morning of the study visit and to bring their medications to the visit with them.
Time Frame: From Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Dapagliflozin 10 mg
Number analyzed (Participants) | 263 | 267
mm Hg | -5.53 (0.8458) | -6.15 (0.8353)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; ANCOVA — Endpoint tested following a sequential testing procedure at 2-sided alpha=0.05 to control the family-wise Type I error rate related to primary and secondary efficacy endpoints. Test not performed since previous tests were not significant; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.96 to 0.73], Standard Error of Mean 0.6866

6. Secondary Outcome: Adjusted Mean Change From Baseline in Serum Uric Acid Levels at Week 12
Description: Central laboratory serum uric acid levels will be determined at the Enrollment, Day -28, Day 1, and at Week 4, 8, 12, and 13 visits. All randomized participants who received at least 1 dose of study drug and who had nonmissing baseline and at least 1 postbaseline value during the double-blind treatment period were used for analysis.
Time Frame: From Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin 10 mg
Number analyzed (Participants) | 279 | 278
mg/dL | 0.05 (0.0747) | -0.27 (0.0754)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Change from baseline to week 12 was calculated using a longitudinal repeated measures analysis using direct likelihood with fixed categorical effects of treatment, week, treatment-by-week interaction, and randomization strata and continuous fixed covariates of baseline value and baseline value by week interaction; Test type: Superiority or Other; Longitudinal repeated measures analysis — Endpoint tested following a sequential testing procedure at two-sided alpha=0.05 to control the family-wise Type I error rate related to primary and secondary efficacy endpoints. Test not performed since previous tests were not significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.46 to -0.18], Standard Error of Mean 0.0717

ADVERSE EVENTS:
Arm/Group | Placebo | Dapagliflozin, 2.5 mg (Randomized Before Protocol Amendment 8) | Dapagliflozin, 5 mg (Randomized Before Protocol Amendment 8) | Dapagliflozin 10 mg
Serious Adverse Events (participants affected / at risk) | 4/311 | 3/166 | 2/165 | 2/302
Other Adverse Events (participants affected / at risk) | 0/311 | 0/166 | 0/165 | 0/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=311) | Dapagliflozin, 2.5 mg (Randomized Before Protocol Amendment 8) (N=166) | Dapagliflozin, 5 mg (Randomized Before Protocol Amendment 8) (N=165) | Dapagliflozin 10 mg (N=302)
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 1 | 0 | 0 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Study originally had 2 additional arms, dapagliflozin 2.5 and 5 mg, but enrolment stopped after Protocol Amendment 8 (1-11-11) implemented. Because endpoints focused on comparison of dapagliflozin 10 mg with placebo, only these arms were summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.